CLINICAL TRIAL: NCT05275504
Title: A Phase I, First-In-Human, Multicenter, Open Label, and Dose-Escalation Study of TT-01488, Administered Orally in Adult Patients With B-Cell Malignancies
Brief Title: Study to Evaluate the Safety and Tolerability of TT-01488 in Patients With B-Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TT01488US01
Record Dates: First submitted 2022-02-21; First posted 2022-03-11 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: B-Cell Malignancies
Keywords: B-Cell Malignancies; Non-Hodgkin's Lymphomas (NHL); BTK inhibitor; C481S mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation for TT-01488 (Experimental): TT-01488 tablets will be administered once daily in a 28-day cycle in increasing strength in order to determine the recommended dose for dose expansion.
  Interventions: Drug: TT-01488
- Dose Expansion for TT-01488 (Experimental): TT-01488 tablets will be administered once daily in 28-day cycles to verify the safety and preliminary efficacy as observed in the dose escalation cohorts.
  Interventions: Drug: TT-01488

INTERVENTIONS:
Drug: TT-01488 — TT-01488 tablet will be administered orally once daily per protocol defined schedule.

SUMMARY:
This is a first-in-human (FIH), multicenter, open-label Phase I dose escalation study to evaluate the safety and preliminary efficacy of the TT-01488 tablet, a non-covalent reversible BTK inhibitor, for the treatment of adult patients with B-cell malignancies.

DETAILED DESCRIPTION:
The study will consist of two parts, dose escalation and dose expansion. A modified 3+3 design will be used to guide the dose escalation and the determination of the dose recommended for dose expansion (DRDE). A sentinel cohort comprising of one subject will be enrolled at a starting dose of 50 mg q.d. Subsequently, patients will be enrolled according to the standard 3+3 dose escalation design to determine the DRDE. Once the DRDE has been selected, TT-01488 of DRDE will be further tested in the dose expansion cohort to verify the safety and preliminary efficacy as observed in the dose escalation cohorts. A recommended Phase II dose (RP2D) may be determined based on the totality of safety, pharmacokinetics, and efficacy data from the dose escalation cohorts and dose expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age with histologically or cytologically confirmed R/R B-NHL, including but not limited to chronic lymphocytic leukemia/small lymphocytic leukemia (CLL/SLL), Waldenström macroglobulinemia (WM), follicular lymphoma (FL), marginal zone lymphoma (MZL), diffuse large-b-cell lymphomas (DLBCL), and transformed lymphoma who failed or are intolerant to ≥ 1 prior standard of care regimens.

   Notes:
   * Patients with prior treatment of BTK inhibitors are eligible
   * Patients with low grade lymphoma must be progressing and requiring treatment:
   * Patients with CLL must have disease requiring treatment as specified in 2018 IWCLL Guidelines (Appendix 5)
   * Patients with B-cell NHL must have measurable disease per 2014 Lugano Classification (Appendix 6)
   * Patients with WM must have minimum serum immunoglobulin M (IgM) level of ≥ 2 times the upper limit of normal (ULN)
2. Body weight ≥ 40 kg
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
4. Adequate organ function, defined by the following laboratory parameters:

   * Hematologic:

     * Absolute neutrophil count (ANC) ≥ 750/ul, unless due to bone marrow involvement due to disease
     * Platelets ≥ 50,000/ul without transfusion within 7 days
     * Hemoglobin ≥ 80 mg/dl without transfusion within 7 days
   * Coagulation:

     * Prothrombin time (PT) ≤ 1.5 × ULN
     * Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
   * Renal function:

     o Creatinine clearance ≥ 60 mL/min estimated glomerular filtration rate based on Cockcroft-Gault formula or 24-hour urine collection
   * Liver function:

     * Total bilirubin ≤ 1.5 × ULN (unless due to Gilbert's disease)
     * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 × ULN unless disease-related
5. Agreement to use contraception during the study and until at least 6 months after the last dose of study drug if sexually active and able to bear children
6. Willing and able to participate in all required evaluations and procedures in the study protocol including swallowing tablets without difficulty
7. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease-free for at least 2 years or which will not limit survival to < 2 years (Note: these cases must be discussed with the Medical Monitor and/or Investigator)
3. A life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of TT-01488, or put the study outcomes at undue risk
4. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or significant screening ECG abnormalities including left bundle branch block, 2nd degree AV block type II, 3rd degree block, bradycardia, and corrected QT interval using Fridericia's Formula (QTcF) > 470 msec, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
5. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
6. Any immunotherapy, , radiotherapy (limited-field radiation for palliation within 7 days), or experimental therapy within 4 weeks, or 5-half lives for chemotherapy and small molecule agents (whichever is shorter), before first dose of study drug (corticosteroids for disease-related symptoms allowed but require 1-week washout before study drug administration)
7. History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor-modified T-cell (CAR-T) therapy within the past 60 days or with any of the following:

   * Active graft versus host disease (GvHD);
   * Cytopenias from incomplete blood cell count recovery post-transplant;
   * Need for anti-cytokine therapy for toxicity from CAR-T therapy; residual symptoms of neurotoxicity > Grade 1 from CAR-T therapy;
   * Ongoing immunosuppressive therapy
8. Concomitant use of prohibited medications(Section 6.4.2), including:

   * Therapeutic doses of warfarin sodium (Coumadin®) or any other coumarin-derivative anticoagulants
   * Medications with known risk to cause QT prolongation or Torsades de pointes
   * Strong CYP3A inhibitors and inducers (must be discontinued for at least 14 days or 5 half-lives, whichever is longer, before study treatment)
   * Proton pump inhibitors, histamine-2 blockers (H2 blockers), and locally acting antacids (Note: For patients who are dependent upon this class of medications, patients may be considered after consulting with the study investigator and Sponsor. See Section 6.4.2 for more details).
9. Central nervous system involvement by lymphoma
10. Grade ≥ 2 toxicity (other than alopecia) continuing from prior anticancer therapy, including radiation
11. Known history of Human Immunodeficiency Virus (HIV) or active infection with Cytomegalovirus (CMV), Hepatitis C Virus (HCV) or Hepatitis B Virus (HBV), or any uncontrolled active systemic infection
12. Major surgery within 4 weeks before first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) of TT-01488 | Up to 28 days after first dose
  Safety and tolerability of TT-01488 as a single agent
Dose recommend for dose expansion (DRDE) | 1 - 1.5 years
  Safety and tolerability of TT-01488 as a single agent
Maximum Tolerated Dose (MTD), if reached, of TT-01488 | Up to 28 days after first dose
  Safety and tolerability of TT-01488 as a single agent

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) | 1 - 1.5 years
  Safety and tolerability of TT-01488 as a single agent. AEs will be assessed per CTCAE v5.0 and may include, but is not limited to, clinically abnormal laboratory tests, physical exams, vital signs, electrocardiograms, and ECOG performance status.
Objective Response Rate (ORR) | 1 - 1.5 years
  Preliminary efficacy profile of TT-01488 as a single agent
Disease Control Rate (DCR) | 1 - 1.5 years
  Preliminary efficacy profile of TT-01488 as a single agent
Duration of Response (DOR) | 1 - 1.5 years
  Preliminary efficacy profile of TT-01488 as a single agent
Progression free survival (PFS) | 1 - 1.5 years
  Preliminary efficacy profile of TT-01488 as a single agent
Overall survival (OS) | 1 - 1.5 years
  Preliminary efficacy profile of TT-01488 as a single agent
Recommended Phase 2 dose (RP2D) | 1 - 1.5 years
  Safety and tolerability of TT-01488 as a single agent
Area under the concentration time curve (AUC 0-last) | 1 - 1.5 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Maximum plasma concentration (Cmax) | 1 - 1.5 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Time to Maximum Plasma Concentration (Tmax) | 1 - 1.5 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Half-life (T1/2) | 1 - 1.5 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Mean Residence Time (MRT) | 1 - 1.5 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent
Volume of Distribution (Vd) | 1 - 1.5 years
  Pharmacokinetic (PK) profile of TT-01488 as a single agent

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, MD, Principal Investigator — The University of Texas MD Anderson Cancer Center (MDACC)
Locations (2):
- United States (2):
  - Gabrail Cancer Center, Canton, Ohio
  - The University of Texas MD Anderson Cancer Center (MDACC), Houston, Texas

IPD SHARING:
Plan to Share IPD: No